CLINICAL TRIAL: NCT04752722
Title: A Phase 1/2 Study of EG-70 as an Intravesical Administration to Patients With BCG Unresponsive Non-Muscle Invasive Bladder Cancer (NMIBC) and High-Risk NMIBC Patients Who Are BCG Naïve or Received Incomplete BCG Treatment
Brief Title: LEGEND Study: EG-70 in NMIBC Patients BCG-Unresponsive and High-Risk NMIBC Incompletely Treated With BCG or BCG-Naïve
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: enGene, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EG-70-101
Record Dates: First submitted 2021-02-04; First posted 2021-02-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Superficial Bladder Cancer; Non-muscle Invasive Bladder Cancer With Carcinoma in Situ
Keywords: Non-muscle invasive bladder cancer (NMIBC); Bacillus calmette- guerin (BCG) failure; BCG unresponsive; NMIBC; Bladder Cancer; LEGEND Study; EG-70; High-risk NMIBC; BCG-naïve; Incomplete BCG treatment; Carcinoma in situ (Cis); BCG-exposed
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Carcinoma in Situ | interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): Dose escalation phase
  Interventions: Drug: EG-70 (phase 1)
- Phase 2 (Experimental): Cohort 1: Recommended Phase 2 dose (RP2D) with eligible BCG-unresponsive NMIBC patients with CIS, up to 4 cycles of treatment with EG-70
  Cohorts 2A, 2B and 3: RP2D with eligible high-risk NMIBC patients with CIS who are BCG-naïve, BCG-exposed (incompletely treated with BCG) or BCG-unresponsive HG Ta/T1 papillary disease without CIS
  Interventions: Drug: EG-70 (phase 2)

INTERVENTIONS:
Drug: EG-70 (phase 1) — Patients will receive up to four cycles of EG-70 administered as a bladder instillation of a 50 mL volume of study drug via catheter with a targeted retention time of 60 minutes.One cycle lasts approximately 12 weeks and consists of either a 2-dose (Day 1 and Day 8) or 4-dose (Day 1, Day 8, Day 29 and Day 36) regimen.
  Other Names: Phase 1
  Arms: Phase 1
Drug: EG-70 (phase 2) — Patients will receive during Treatment Period, up to 4 cycles of EG-70 at the RP2D defined in Phase 1 administered as a bladder instillation of a 50 mL volume of study drug via catheter with a targeted retention time of 60 minutes. One cycle lasts approximately 12 weeks. For Maintenance treatment 2 doses of EG-70 will be administered as a bladder instillation per 12-week cycle.
  Other Names: Phase 2
  Arms: Phase 2

SUMMARY:
This study will evaluate the safety and efficacy of intravesical administration of EG-70 in the bladder and its effect on bladder tumors in patients with NMIBC.

This study study consists of two phases; a Phase 1 dose-escalation to establish safety and recommended the phase 2 dose, followed by a Phase 2 study to establish how effective the treatment is.

The Study will include patients with NMIBC with Cis for whom BCG therapy is unresponsive and patients with NMIBC with Cis who are BCG-naïve or inadequately treated.

DETAILED DESCRIPTION:
EG-70 is a novel non-viral gene therapy. EG-70 is designed to elicit a local immune response following delivery of the study gene therapy to the bladder urothelium. This approach of local administration through bladder instillation has the potential to induce a potent immune response exclusively at the site of the tumor, resulting in greater therapeutic benefit while reducing undesirable systemic toxicity.

Eligible BCG-unresponsive NMIBC patients will be enrolled in Phase 1, and Cohort 1 of Phase 2.

Eligible high-risk NMIBC patients will be enrolled starting in Phase 2 in separate single are cohorts include: BCG-naïve patients or BCG-exposed (incompletely treated) patients with Carcinoma in situ (CIS), and BCG-unresponsive HG Ta/T1 papillary disease without CIS.

Patients will be treated for up to four 12-week cycles of study drug instillation doses and assessments with follow up assessments.

Patients with complete response following the four 12-week cycles will enter up to 4 maintenance treatment cycles, and those remaining in complete response will enter another 4 maintenance treatment cycles or follow up assessments.

ELIGIBILITY:
Inclusion Criteria:

BCG-unresponsive Patients:

1. BCG-unresponsive NMIBC with carcinoma in situ (CIS) with or without coexisting papillary Ta/T1 tumors who are ineligible for or have elected not to undergo cystectomy, and have experienced CIS disease within 12 months of treatment where: adequate BCG regimen consists of at least 2 courses of BCG where the first course (induction) must have included at least 5 or 6 doses and the second course may have included a re-induction (at least 2 treatments) or maintenance (at least 2 doses), and Cis must be documented or indicated by pathology

   Phase 2 Only:
2. BCG-Naïve or BCG-incompletely treated Patients with CIS or BCG-unresponsive, HG Ta/T1 papillary disease without CIS:

   -NMIBC with current Cis of the bladder, with or without coexisting papillary Ta/T1 NMIBC tumor(s), who are ineligible for or have elected not to undergo cystectomy, where: either: cohort 2a) no treatment with BCG but may have previously been treated with at least 1 dose of intravesical chemotherapy following transurethral resection of bladder tumor (TURBT) and Cis must be documented or cohort 2b) indicated by pathology incomplete BCG treatment (at least 1 dose and less than the 5+2 doses required for adequate dosing per Cohort 1) or cohort 3) patients who are BCG-unresponsive following adequate treatment, with HG Ta/T1 papillary disease without CIS.

   All Patients:
3. Patients who have previously been treated with a checkpoint inhibitor and failed treatment are eligible for inclusion 30 days post-treatment (Phase 1) or 3 months post-treatment (Phase 2).
4. Male or non-pregnant, non-lactating female, 18 years or older.
5. Women of childbearing potential must have a negative pregnancy test at Screening.
6. Female patients of childbearing potential must be willing to consent to using highly effective birth control methods; Male patients are required to utilize a condom for the duration of the study treatment through 3 months post-dose.
7. In Phase 2, for patients with T1 lesions may be eligible after repeat TURBT if pathology shows non-invasive (Ta or less) or no disease.
8. Performance Status: Eastern Cooperative Oncology Group 0, 1, and 2.
9. Hematologic inclusion: a. Absolute neutrophil count >1,500/mm3. b. Hemoglobin >9.0 g/dL. c. Platelet count >100,000/mm3.
10. Hepatic inclusion: a. Total bilirubin must be ≤1.5 x the upper limit of normal (ULN). b. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase ≤2.5 x ULN.
11. Adequate renal function with creatinine clearance >30 mL/min
12. Prothrombin time and partial thromboplastin time ≤1.25 x ULN or within the therapeutic range if on anticoagulation therapy.
13. Must have satisfactory bladder function with ability to retain study drug for 60 minutes.

Exclusion Criteria:

1. Active malignancies (i.e., progressing or requiring treatment change in the last 24 months). Exceptions allowed under Sponsor review.
2. Concurrent treatment with any chemotherapeutic agent.
3. History of partial cystectomy.
4. Treatment with last therapeutic agent (including intravesical chemotherapy post-TURBT) within 30 days of Screening (prior to the screening biopsy).
5. Patients who have received systemic immunosuppressive medication including high-dose corticosteroids.
6. History of severe asthma or other respiratory diseases.
7. History of unresolved vesicoureteral reflux or an indwelling urinary stent.
8. History of unresolved hydronephrosis due to ureteral obstruction.
9. Participation in any other research protocol involving administration of an investigational agent within 30 Days prior to screening or any prior treatment of NMIBC with any investigational gene or immunotherapy agent.
10. History of external beam radiation to the pelvis or prostate brachytherapy within the last 12 months.
11. History of interstitial lung disease and/or pneumonitis in patients who have previously received a PD-1 or PD-L1 inhibitor therapy.
12. Evidence of metastatic disease.
13. History of difficult catheterization that in the opinion of the Investigator will prevent administration of EG-70.
14. Active interstitial cystitis on cystoscopy or biopsy.
15. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
16. Known human immunodeficiency virus, Hepatitis B, or Hepatitis C infection.
17. Significant cardiovascular risk (e.g., coronary stenting within 8 weeks, myocardial infarction within 6 months).
18. Hypersensitivity to any of the excipients of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Nature, incidence, relatedness, and severity of all AEs and SAEs according to the CTCAE v5.0. | Approximately 2 years
  The type, incidence, relatedness and severity of treatment emergent adverse events of EG-70 as assessed by NCI-CTCAE V5.0 will be monitored.
Phase 2: Percentage of patients with cystoscopic CR at 48 weeks, based on exam, urine cytology and appropriate biopsies. | Approximately 48 weeks
  Complete response rate will be measured by determining the number of patients without recurrence of high-grade disease.
Phase 2: Nature, incidence, relatedness, and severity of treatment emergent adverse events (as assessed by CTCAE v5.0) | Approximately 3 years
  The type, incidence, relatedness and severity of treatment emergent adverse events of EG-70 as assessed by NCI-CTCAE V5.0 will be monitored.

SECONDARY OUTCOMES:
Phase 1: The number of patients who experience a DLT through the end of Cycle 1 | Approximately 12 Weeks
  To identify the number of patients who experience a DLT through the end of Cycle 1
Phase 1: CR rate to EG-70 by cystoscopy at approximately 12 weeks. | Approximately 12 weeks
  To evaluate preliminary efficacy of EG-70 by 12 weeks via cystoscopy
Phase 2: Progression-free survival (PFS) | Approximately 3 years
  To evaluate disease-free survival rate
Phase 2: CR rate at 12, 24, 36, and 96 weeks | Approximately 12, 24, 36, and 96 weeks
  To further evaluate CR at the efficacy analysis following each cycle.
Phase 2: Duration of response of the responding patients | Approximately 3 years
  Durability will be measured by determining the number of patients without recurrence of high-grade disease.
Phase 2: Quality of Life Assessment | 24 weeks
  Health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Christine Tosone, Ms, RAC, Study Director — enGene, Inc.
Locations (100):
- United States (49):
  - The University of Alabama at Birmingham Clinical Research Unit (CRU), Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - Urological Associates of South Arizona, Tucson, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - University of California - Irvine Medical Center, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Tower Urology, Los Angeles, California
  - Genesis Research, San Diego, California
  - Colorado Clinical Research, Lakewood, Colorado
  - The George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Florida, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center / University of Miami Hospital and Clinics, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Urology of Indiana, Greenwood, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - John Hopkins Hospital, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Corewell Health Medical Group and Spectrum Health Hospitals, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New Jersey Urology, LLC, Voorhees Township, New Jersey
  - Albany Medical College, Albany, New York
  - Mount Sinai Medical Center, New Haven, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Associated Medical Professionals of NY,, Syracuse, New York
  - UNC Chapel Hill Hospital, Chapel Hill, North Carolina
  - Duke Health - Duke Cancer Center, Durham, North Carolina
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Central Ohio Urology Group, Gahanna, Ohio
  - Clinical Research Solutions - Helios Clinical Research, Middleburg Heights, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - Vanderbilt Univerity Medical Center, Nashville, Tennessee
  - Urology Austin, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Metro Urology, Houston, Texas
  - Houston Methodist Hospital - Department of Urology, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - Froedtert Hospital / Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - Icon Cancer Center Windsor Gardens, Windsor Gardens, South Australia
- Canada (6):
  - Prostate Cancer Centre, Calgary, Alberta
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Center - Glen site, Montreal, Quebec
  - CHUM Centre Hospitalier de l Universite de Montreal, Montreal, Quebec
- France (7):
  - CHU d'Angers, Angers
  - CHU Bordeaux Pellegrin, Bordeaux
  - lnstitut Bergonie 229 Cour de l'Argonne, Bordeaux
  - CHU de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Hopital Bichat Claude-Bernard, Paris
  - CHU de Rauen- Hopital Charles Nicolle, Rouen
- Germany (6):
  - Klinik fur Urologie, Uro-Onkologie, spezielle urologische und Roboter-assistierte Chirurgie Universitatsklinikum Koln (AOR), Cologne
  - Urologicum Duisburg, Duisburg
  - Universitaetsklinikum Erlangen, Erlangen
  - Urologie Neandertal Mettmann, Mettmann
  - Studienpraxis Urologie, Nürtingen
  - Universitaetsklinikum Tubingen, Tübingen
- Italy (6):
  - Clinic Unit of Urology, IRCCS Ospedale San Raffaele, Milan, MI
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Fondazione Policlinico Universitario "A.Gemelli" IRCCS, Largo, Rome
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Rome
  - UOC Urologia, IFO- lstituto Tumori "Regina Elena", Rome
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam, Gyunggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Soul St. Mary's Hospital, Seoul
- Spain (12):
  - IOB - Hospital Quironsalud Barcelona, Barbera Del Valles
  - Fundacio Puigvert, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Quironsalud Madrid (Next Oncology), Madrid
  - Hospital Universitario Infanta Sofia, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Marqués de Valdecilla,, Santander
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No